CLINICAL TRIAL: NCT07055022
Title: Low-level Light Therapy Versus Intense Pulsed Light to Prevent Iatrogenic Dry Eye Disease After Cataract Surgery: a Randomised Controlled Trial
Brief Title: Low-level Light Therapy Versus Intense Pulsed Light to Prevent Iatrogenic Dry Eye Disease After Cataract Surgery
Acronym: EDACS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Trenel (Other)
Collaborators: ProSurg (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025-A00858-41
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Cataract Surgery; Eye Dryness
Keywords: IPL; LLLT; Intense Pulse Light; Low Level Light Therapy; cataract surgery; phacoemulsification; prophylaxis; prevention; eye dryness; dry eye disease; DED
MeSH Terms: conditions — Xerophthalmia; Dry Eye Syndromes | interventions — Low-Level Light Therapy; Phototherapy; Intense Pulsed Light Therapy

STUDY DESIGN:
Intervention Model Description: A randomised controlled surgeon-blinded, evaluator-blinded monocentric trial in a non-inferiority framework with a 1:1 allocation ratio.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Surgeons and the medical staff (the evaluators) that administer the questionnaires will be blinded to the randomisation, but the orthoptists performing the treatment will be aware of the randomisation. Participants will not be informed of their allocated treatment; however, they may guess which treatment they received as the IPL and LLLT devices look differently, and the patient can see the device being used. Moreover, the patient's experience will be different. In the IPL group, light is administered in pulses and the patients experience heat; furthermore, cooling ultrasound gel and eye patches are used for protection. In the LLLT group, light is administered continuously, and there is no protective gel nor eye patches. At the end of the study, participants may request what type of treatment they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPL (Active Comparator): Patients in the IPL group will receive 3 sessions of IPL treatment with OptiClear device (Alma Lasers GmbH, Nuremberg, Germany) at D-7, D+7, and D+30. Each session will comprise 90 homogenously spaced pulses of light (wavelength of 550-650 nm, pulse time 10,12 or 15 ms, pulse repetition rate 1-2 Hz) using an energy density of 8-12 J/cm2 adjusted to Fitzpatrick skin type according to the manufacturer's recommendations. The treatment will be applied to the lower eyelid region. Ultrasound gel, as well as protective eye patches will be used, and the patients will be asked to close their eyes during the session. The chosen parameters are currently used in the clinical practice of the participating surgeons as treatment for DED; moreover, similar values are reported in published studies
  Interventions: Procedure: IPL
- LLLT (Experimental): Patients in the LLLT group will receive 3 sessions of LLLT treatment with Eye-light device (Espansione Group S.p.A., Bologna, Italy) 7 days before phacoemulsification (D-7), 7 days after phacoemulsification (D+7), and 30 days after phacoemulsification (D+30). Each session will consist of 15 minutes of light treatment using a wavelength of 625±40 nm and maximum power of 10 W (maximal total fluence of 32 J/cm2 ± 20% per session) applied on the periorbital region. The patients will be asked to close their eyes during the session. The chosen parameters are currently used in the clinical practice of the participating surgeons as treatment for DED; moreover, similar values are reported in published studies
  Interventions: Procedure: LLLT

INTERVENTIONS:
Procedure: LLLT — Patients in the LLLT group will receive 3 sessions of LLLT treatment with Eye-light device (Espansione Group S.p.A., Bologna, Italy) 7 days before phacoemulsification (D-7), 7 days after phacoemulsification (D+7), and 30 days after phacoemulsification (D+30). Each session will consist of 15 minutes of light treatment using a wavelength of 625±40 nm and maximum power of 10 W (maximal total fluence of 32 J/cm2 ± 20% per session) applied on the periorbital region. The patients will be asked to close their eyes during the session. The chosen parameters are currently used in the clinical practice of the participating surgeons as treatment for DED; moreover, similar values are reported in published studies
  Other Names: Low Level Light Therapy; phototherapy; photobiomodulation; cold laser therapy
  Arms: LLLT
Procedure: IPL — Patients in the IPL group will receive 3 sessions of IPL treatment with OptiClear device (Alma Lasers GmbH, Nuremberg, Germany) at D-7, D+7, and D+30. Each session will comprise 90 homogenously spaced pulses of light (wavelength of 550-650 nm, pulse time 10,12 or 15 ms, pulse repetition rate 1-2 Hz) using an energy density of 8-12 J/cm2 adjusted to Fitzpatrick skin type according to the manufacturer's recommendations. The treatment will be applied to the lower eyelid region. Ultrasound gel, as well as protective eye patches will be used, and the patients will be asked to close their eyes during the session. The chosen parameters are currently used in the clinical practice of the participating surgeons as treatment for DED; moreover, similar values are reported in published studies
  Other Names: Intense Pulsed Light
  Arms: IPL

SUMMARY:
Dry eye disease (DED) is a frequent ocular surface disease (OSD) of multifactorial origin, characterised by disruption of tear film homeostasis and associated with ocular discomfort and/or visual disturbance. Cataract surgery, which is one of the most often performed interventions worldwide, can induce or worsen the symptoms of DED. Despite lack of guidelines on DED prophylaxis before cataract surgery in the general population, there is a growing interest in this topic due to the high prevalence of postoperative DED. A recent randomised controlled trial (RCT) with one month follow-up showed that prophylactic low-level light therapy (LLLT) before and after cataract surgery in patients without pre-existing DED significantly improved postoperative tear film stability, as well as reduced ocular discomfort, compared to no prophylaxis. Apart from LLLT, another light-based treatment for DED is intense pulsed light (IPL); the treatments have shown favourable outcomes in the management of DED, both as stand-alone choices or in combination.

DETAILED DESCRIPTION:
Dry eye disease (DED) is a frequent ocular surface disease (OSD) of multifactorial origin, characterised by disruption of tear film homeostasis and associated with ocular discomfort and/or visual disturbance. Cataract surgery, which is one of the most often performed interventions worldwide, can induce or worsen the symptoms of DED. Despite lack of guidelines on DED prophylaxis before cataract surgery in the general population, there is a growing interest in this topic due to the high prevalence of postoperative DED. A recent randomised controlled trial (RCT) with one month follow-up showed that prophylactic low-level light therapy (LLLT) before and after cataract surgery in patients without pre-existing DED significantly improved postoperative tear film stability, as well as reduced ocular discomfort, compared to no prophylaxis. Apart from LLLT, another light-based treatment for DED is intense pulsed light (IPL); the treatments have shown favourable outcomes in the management of DED, both as stand-alone choices or in combination.

There is currently no comparative data available which would allow to choose between LLLT and IPL as prophylaxis for iatrogenic DED after cataract surgery.

The primary objective of this RCT is to compare LLLT versus IPL as prophylaxis for iatrogenic DED after cataract surgery in terms of patient-reported symptoms of eye dryness at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥50 years
* scheduled for bilateral cataract surgery by phacoemulsification
* without current DED treatment, including eye drops, for at least two months before the inclusion
* with preoperative OSDI ≤22 points, indicating absence of DED or mild DED
* who signed the informed consent and are willing to comply with the protocol requirements based on the investigator's judgment
* affiliated with a social security scheme
* with an ability to answer questionnaires and to communicate freely in French.

Exclusion Criteria:

* set to undergo implantation of a multifocal intraocular lens
* using contact lenses
* with any of the following in the included eye: (i) age-related macular degeneration (AMD), (ii) previous ocular surgery, (iii) abnormal clinical exam of the ocular surface or (iv) undergoing any ocular treatment
* with systemic contraindications, including autoimmune diseases (e.g., Sjögren syndrome)
* with general contraindications for LLLT or IPL treatment: dark pigmented skin (Fitzpatrick grade ≥5), skin photosensitivity (regardless if innate, pathological or medically-induced), or neurological light sensitivity (e.g. epilepsy, light-induced migraines)
* with contraindications for LLLT or IPL treatment limited to the treatment area: history of skin cancer, skin pigmented lesions, as well as fixed/permanent skin piercings, face tattoos, semi-permanent make-up (including microblading) or skin defects
* with any concomitant disease or disorder which, in the opinion of the investigator, may put the patient at risk or may influence the result of the study
* with protected status under articles L1121-6, LL121-8 and L1122-2 of the French Public Health Code
* who cannot comply with the protocol requirements based on the investigator's judgment.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient-reported symptoms of eye dryness (OSDI) | 3 months after cataract surgery
  Participants will be asked to report the symptoms of eye dryness by answering an OSDI questionnaire assisted by a member of the medical staff (blinded to the randomisation). OSDI is a widely used, validated questionnaire for the diagnosis of DED and evaluation of its severity and consists of 12 items graded from 0 (never) to 4 (all the time). The final OSDI score is within the range of 0 (no disability) to 100 (complete disability) and is calculated based on the following formula: [(sum of scores for the questions answered) × 25] / (total number of questions answered).

SECONDARY OUTCOMES:
Patient-reported symptoms of eye dryness (OSDI) | 1 week, 1 month after cataract surgery
  Participants will be asked to report the symptoms of eye dryness by answering an OSDI questionnaire assisted by a member of the medical staff (blinded to the randomisation). OSDI is a widely used, validated questionnaire for the diagnosis of DED and evaluation of its severity and consists of 12 items graded from 0 (never) to 4 (all the time). The final OSDI score is within the range of 0 (no disability) to 100 (complete disability) and is calculated based on the following formula: [(sum of scores for the questions answered) × 25] / (total number of questions answered).
patient-reported symptoms of eye dryness (SANDE) | 1 week after, 1 month after and 3 months after the surgery
  Participants will answer a Symptom Assessment in Dry Eye (SANDE) questionnaire assisted by a member of the medical staff (blinded to the randomisation). SANDE consists of two questions: "How often, on average, do your eyes feel dry and/or irritated?" and "How severe, on average, do you feel your symptoms of dryness and/or irritation are?". The patient answers both of them on a 100-mm horizontal visual analogue scale (VAS). The location of the mark made by the patient for each question is measured in mm from the left-hand side of the 100-mm line. The final score is calculated by multiplying frequency and severity scores and calculating the square root of the result
Non-invasive tear film break-up time (NIBUT) | 1 week, 1 and 3 months after cataract surgery
  Automated corneal surface analysis using CA-900 corneal topographer (Topcon Healthcare, Tokyo, Japan)
Ocular redness | 1 week after, 1 and 3 months after cataract surgery
  Automated corneal surface analysis using CA-900 corneal topographer (Topcon Healthcare, Tokyo, Japan), on 0-4 Efron scale, grade 0 corresponding to normal ocular redness; a high quality image is obtained with CA-900 and Efron scale is displayed on the screen for a manual comparison
Meibomian gland (MG) atrophy | 1 week, 1 and 3 months after cataract surgery
  a) Automated corneal surface analysis using CA-900 corneal topographer (Topcon Healthcare, Tokyo, Japan), on 1-4 scale, grade 1 corresponding to <25% of MG atrophy; grade 2: 25% < atrophy < 50%; grade 3: 50% < atrophy < 75%; grade 4: atrophy > 75%
Fluorescein corneal staining (FCS) | 1 week, 1 and 3 months after cataract surgery
  With 0.5% fluorescein (SERB SA, Bruxelles, Belgium) assessed under a slit lamp, on 1-4 scale, grade 1 corresponding to no punctate staining; grade 2: no punctate staining but eye tearing/watering; grade 3: localised punctate staining; grade 4: diffuse punctate staining or staining fused in plaques
Eyelid telangiectasias | 1 week after, 1 and 3 months after cataract surgery
  Assessed under a slit lamp, on 1-4 scale, grade 1 corresponding to no telangiectasias; grade 2: eyelid (skin) or eyelid margin telangiectasias; grade 3: superficial telangiectasias of inferior palpebral conjunctiva; grade 4: deep telangiectasias of inferior palpebral conjunctiva
Meibomian expressiblity and quality | 1 week, 1 and 3 months after cataract surgery,
  Assessed under a slit lamp, on 1-4 scale, grade 1 corresponding to no MG obstruction, clear and easily expressed meibum; grade 2: cloudy meibum of abnormal viscosity; grade 3: thick, toothpaste-like or filament-like meibum, difficult to express; grade 4: MG obstruction with no meibum expression even under significant pressure
Ultrasound energy delivered | Intra-operatively
  Collected during the cataract surgery as cumulative dissipated energy (CDE), obtained as an automatically calculated value displayed at the end of the surgery on the screen of the phacoemulsification system
Adverse Events | 0 to 3 months after cataract surgery
  Including complications and reoperations, specifying the incidence, severity, and relationship to the treatment applied

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Trenel, Sainte-Colombe, France

IPD SHARING:
Plan to Share IPD: No